CLINICAL TRIAL: NCT07252622
Title: Progesterone Levels and Frozen Embryo Transfer Outcomes
Acronym: PLATO
Status: Not yet recruiting | Type: Observational
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00089821
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: IVF
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood draw — All patients will have one additional blood draw on the day of their transfer to measure progesterone level.

SUMMARY:
Frozen embryo transfers (FET) now represent the majority of all embryo transfer cycles, and upwards of 60% live births in United States are now attributable to frozen embryo transfers (1). Exogenous progesterone for endometrial decidualization and luteal phase support is thought to be critical to both optimizing endometrial receptivity for implantation as well as sustaining early pregnancy prior to reliable secretory activity of the early placenta.

The purpose of this study is to:

1. Determine the prevalence of low serum progesterone levels (less than 10 ng/ml) among patients undergoing a programmed embryo transfer cycle on the day of frozen embryo transfer.
2. Determine if serum progesterone < 10 ng/ml on the day of frozen embryo transfer is associated with poorer FET outcomes: ongoing pregnancy (primary outcome), live birth, biochemical pregnancy, and clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Female patient undergoing programmed frozen embryo transfer using exogenous estrogen and progesterone, with exogenous progesterone administered via a combination of vaginal progesterone (Endometrin®) (2-3 times daily) and intermittent progesterone-in-oil (PIO) (every 3rd day) according to standard protocol. Protocols involving other formulations of vaginal progesterone (e.g. Crinone®, Prometrium®, will also be included).
3. Planned transfer one 1 euploid embryo. Recruited patients will have at least 1 euploid embryo available for transfer.
4. Standard eligibility criteria to undergo frozen embryo transfer at Shady Grove Fertility.
5. 18 years and older

Exclusion Criteria:

1. Age less than 18 years or greater than 51 years
2. Planned intervention based on serum progesterone concentration measured any time after initiation of intramuscular or vaginal progesterone.
3. Uterine cavity abnormality that has not been surgically corrected.
4. Any medical or surgical contraindication to undergoing programmed frozen embryo transfer or pregnancy.
5. Planned use of embryos cryopreserved by slow-freeze, prior to blastocyst stage, or other than PGT-A normal.
6. Currently breast feeding, pregnancy, or having a contraindication to pregnancy.
7. Participation in any experimental drug study within 60 days prior to screening.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: All patients undergoing programmed frozen embryo transfer of a single euploid embryo with combined vaginal progesterone and intramuscular PIO.
Sampling Method: Non-Probability Sample
Enrollment: 659 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy | Through study completion, an average of 1 year
  At the completion of the study, a chart review will be performed to determine which patients who participated in this study have an ongoing pregnancy. This information is recorded in our electronic medical record as a binary variable (ongoing pregnancy - yes or no).

IPD SHARING:
Plan to Share IPD: No